CLINICAL TRIAL: NCT05481567
Title: Oral Health Related Quality of Life in Patients Affected by Periodontitis Stage III and IV: a Survey Based on OHIP14 Questionnaire
Brief Title: Periodontitis Stage III and IV and Oral Health Related Quality of Life
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Nicola Alberto Valente, DDS, MS, PhD, Assistant Professor, University of Cagliari
Other Study IDs: Perio3
Record Dates: First submitted 2022-07-25; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Periodontitis
Keywords: Periodontitis; OHIP14; Quality of life; Questionnaire
MeSH Terms: conditions — Periodontitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stage III: Patients diagnosed with periodontitis stage III
  Interventions: Other: Questionnaire
- Stage IV: Patients diagnosed with periodontitis stage IV
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A series of 14 questions about with the impact of periodontitis on quality of life.

SUMMARY:
Patients diagnosed with stage III or IV periodontitis during routine visits at the department of periodontology will undergo a validated questionnaire to understand the impact of the disease on their quality of life.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the impact of stage III and stage IV periodontitis on the quality of life of patients and to evaluate the differences of the results between the two forms of the disease.

Patients who presents to our periodontology department for routine follow-up visits, if diagnosed with one of these two forms of periodontitis, will be asked if they intend to answer a short questionnaire with the intent to understand how the disease affects their daily activities and interactions.

The questionnaire that will be used is the short-form Oral Health Impact Profile (OHIP-14), which consists of 14 questions each one formulated in the following way: "How often (impact item) because of problems with your teeth, mouth, or dentures?" The impact items belong to seven different impact domains: (a) functional limitations, (b) physical pain, (c) psychological discomfort, (d) physical disability, (e) psychological disability, (f) social disability, and (g) handicap. Each question could be answered with a score from 0 to 4 corresponding to: 0 = never, 1 = hardly ever, 2 = occasionally, 3 = fairly often, and 4 = very often.

The impact items are:

Had trouble in pronouncing words Felt that sense of taste had worsened Had painful aching in your mouth Found it uncomfortable when eating food Been feeling self-conscious Have you felt tense Diet has been unsatisfactory Had to interrupt meals Found it difficult to relax Been a bit embarrassed Been irritable with other people Had difficulty during usual jobs Felt that life less satisfying Been totally unable to function Overall mean scores as well as for each question and for each impact domain will be calculated and compared with two ways ANOVA statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by periodontitis stage III
* Patients affected by periodontitis stage IV

Exclusion Criteria:

* Patients affected by periodontitis stage I
* Patients affected by periodontitis stage II

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any age affected by periodontitis stage III or stage IV willing to answer a questionnaire about their quality of life
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall score | 1 day (At the time of evaluation, the first time the patients is evaluated and diagnosed with either periodontitis stage III or stage IV)
  The sum of the scores of each of the seven impact domains of the Oral Health Impact Profile OHIP14 survey (0 = never to 4 = very often)

SECONDARY OUTCOMES:
Impact domain score | 1 day (At the time of evaluation, the first time the patients is evaluated and diagnosed with either periodontitis stage III or stage IV)
  The sum of the scores of each of the seven impact domains of the Oral Health Impact Profile OHIP14 survey (0 = never to 4 = very often)

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Duilio Casula, AOU Cagliari, Monserrato, CA, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared in a publication after the end of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be submitted for publication right after the analysis of the outcomes

REFERENCES:
- [Background] Palaiologou A, Kotsakis GA. Dentist-Patient Communication of Treatment Outcomes in Periodontal Practice: A Need for Dental Patient-Reported Outcomes. J Evid Based Dent Pract. 2020 Jun;20(2):101443. doi: 10.1016/j.jebdp.2020.101443. Epub 2020 Apr 27. PMID 32473794
- [Result] Khan S, Khalid T, Bettiol S, Crocombe LA. Non-surgical periodontal therapy effectively improves patient-reported outcomes: A systematic review. Int J Dent Hyg. 2021 Feb;19(1):18-28. doi: 10.1111/idh.12450. Epub 2020 Jul 16. PMID 32594621
- [Result] Sharma P, Yonel Z, Busby M, Chapple IL, Dietrich T. Association between periodontal health status and patient-reported outcomes in patients managed in a non-specialist, general dental practice. J Clin Periodontol. 2018 Dec;45(12):1440-1447. doi: 10.1111/jcpe.13022. Epub 2018 Nov 5. PMID 30341963
- [Result] Baiju RM, Peter E, Varghese NO, Anju P. Patient Reported Outcome Assessment of Periodontal Therapy: A Systematic Review. J Clin Diagn Res. 2017 Aug;11(8):ZC14-ZC19. doi: 10.7860/JCDR/2017/28505.10343. Epub 2017 Aug 1. PMID 28969266